CLINICAL TRIAL: NCT02926144
Title: Can the Use of the McGRATH® MAC Videolaryngoscope Decrease the Number of People Required for Tracheal Intubation in a Population of Patients Without Predicted Difficult Intubation?
Brief Title: Does McGRATH® MAC Videolaryngoscope Decrease the Number of People Required to Perform Intubation During Anesthesia ?
Acronym: MGM3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016/05; 2016-A00056-45 (Other: ANSM)
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Anesthesia
Keywords: Intratracheal intubation; videolaryngoscope; McGrath MAC
MeSH Terms: interventions — Laryngoscopes; Intubation, Intratracheal; Intubation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laryngoscope with video (Experimental): Use of the video-laryngoscope McGrath Mac with use of the video feature
  Interventions: Device: Laryngoscope with video
- Laryngoscope without video (Active Comparator): Use of the video-laryngoscope McGrath Mac without use of the video feature
  Interventions: Device: Laryngoscope without video

INTERVENTIONS:
Device: Laryngoscope with video — Intubation with video-laryngoscope McGrath with use of the video feature
  Other Names: Endotracheal intubation with laryngoscope video feature
  Arms: Laryngoscope with video
Device: Laryngoscope without video — Endotracheal intubation with video-laryngoscope McGrath without use of the video feature
  Other Names: Intubation without the laryngoscope video feature
  Arms: Laryngoscope without video

SUMMARY:
The main objective of this study is to compare the proportion of tracheal intubations for which more than one person is necessary when using the McGRATH® MAC videolaryngoscope.

DETAILED DESCRIPTION:
Videolaryngoscopes, such as McGRATH® MAC videolaryngoscope, are used to facilitate tracheal intubations. This study is designed to evaluate the proportion of cases requiring more than one member of the anesthesiology team when the video feature of McGRATH® MAC is available during laryngoscopy in a population of patients without a predicted difficult intubation (Arne's score <11).

General anesthesia from induction until tracheal intubation is recorded on a video for further analysis. Analysis includes characteristics of intubation, patient's monitoring and cooperation between anesthesiologists in two groups. In the control group, the screen of the McGRATH® MAC videolaryngoscope is hidden. In the experimental group, the McGRATH® MAC videolaryngoscope is used with its video feature.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old minimum
* Requiring general anesthesia and orotracheal intubation with a single lumen tube
* Having signed an inform consent form
* Having a telephone and agreeing to communicate their phone number
* Benefiting from a social insurance scheme or beneficiary

Exclusion Criteria:

* Pregnant or breast-feeding women
* Patients taken care in ambulatory surgery who could not be contacted within 24 hours following surgery
* Patients having a predicted difficult intubation (Arné's score ≥ 11) or predicted difficult mask ventilation
* patients requiring a rapid-sequence intubation
* patients for whom general anesthesia using sufentanil, propofol, atracurium or rocuronium is not suitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Number of people needed for tracheal intubation when the video feature of McGRATH® MAC videolaryngoscope is available | 30 minutes
  Intubation is video and audio recorded for further analysis. The availability of the video feature of McGRATH® MAC is hidden from the recording. Only the number of people required and the intubation characteristics can be seen on the video.

SECONDARY OUTCOMES:
Cooperation between members of the anesthesiology team during intubation | 30 minutes
  Based on the video recording: Use of the Kraus Scale (based on "Kraus M, Huang C, Keltner D: Tactile Communication, Cooperation and Performance. Emotion, 2010, 10, 745-9") evaluating communication and gestures within the team
Intubation difficulty Scale (IDS) | 30 minutes
Number of hands necessary for tracheal intubation | 30 minutes
  Based on the video recording: 2 hands when one person intubates by itself without any help, 3 or 4 hands when assistance is given by a second anesthesiologist. 5 to 6 hands when a third person is needed.
Time to intubate | 30 minutes
  Based on the video recording: from the entrance of the blade in the patient's mouth until the presence of the first capnogram
Esophageal intubation | 30 minutes
  No capnograms during mechanical ventilation once intubation is performed
Intubation failure | 30 minutes
  Based on the video recording
Arterial desaturation | 30 minutes maximum
  Based on the video recording: visualisation of a pulse oximetry inferior to 92%
Perception of intubation difficulty by the operator | 30 minutes
  Evaluation on a scale between zero (no difficulty at all) to ten (extremely difficult)
Impact of videolaryngoscopy on hemodynamic variables | 30 minutes
  Based on the video recording: Blood pressure and heart beat on monitoring before and after video laryngoscopy
Evaluation of usual complications after tracheal intubation | 24 hours
  Sore throat or voice change noticed on day 1

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Belze, MD, Principal Investigator — Hopital Foch
Locations (4):
- France (4):
  - Institut Hospitalier Franco Britannique, Levallois-Perret
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - Centre Clinical, Soyaux
  - Hopital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: Yes
Data will be available in the Dryad repository.
Supporting Information: Analytic Code
Time Frame: After publication in a peer-review journal. No limit in time
Access Criteria: No criteria
URL: https://datadryad.org/stash

REFERENCES:
- [Derived] Belze O, Coppere Z, Ouattara J, Thion LA, Paqueron X, Devys JM, Ma S, Kennel T, Fischler M, Le Guen M. Influence of videolaryngoscopy using McGrath Mac on the need for a helper to perform intubation during general anaesthesia: a multicentre randomised video-no-video trial. BMJ Open. 2022 Jan 3;12(1):e049275. doi: 10.1136/bmjopen-2021-049275. PMID 34980609